CLINICAL TRIAL: NCT01306734
Title: Hypothermia and Circulatory Arrest During Surgery on the Ascending Aorta: A Comparison Between Two Cooling Methods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HYPO-SKS-2011
Record Dates: First submitted 2011-01-07; First posted 2011-03-02 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Ascending Aorta Aneurism
Keywords: Extracorporeal circulation; Deep Hypothermic Circulatory Arrest; aortic aneurism; neurological injury; inflammation; coagulation
MeSH Terms: conditions — Trauma, Nervous System; Inflammation; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gradient cooling group: Study group receiving gradient cooling during the procedure using extracorporeal circulation (ECC). The procedure is used routinely in the department and is not an experimental procedure. A maximum of 10 degrees celsius is allowed between the measured nasopharyngeal body temperature and the heater-cooler unit of the ECC-machine, when cooling or rewarming.
- Crash cooling group: Study group receiving rapid cooling using extracorporeal circulation. The protocol for rapid cooling is using routinely in the department and is not an experimental procedure. When cooling, the investigators aim for maximal difference in temperature between the heater-cooler unit of the ECC-machine.

SUMMARY:
PURPOSE: To compare crash cooling versus gradient cooling methods for patients undergoing planned surgery on the ascending aorta in deep hypothermic circulatory arrest. To investigate the impact of hypothermia and circulatory arrest on the coagulation, stress-response, and cerebral outcome.

BACKGROUND: Cooling to 18 °C using extracorporeal circulation allows for circulatory arrest during surgery on the ascending aorta. Two different methods are used either lowering the temperature of the blood by 10 °C at a time, gradient cooling, or as cold as possible, crash cooling. The distribution of hypothermia is expected to be different for the two methods, the latter predominantly cooling the body core. The influence on the physiological response is expected to vary with the two methods. The surgical procedure and the cooling greatly elicit a stress response and the coagulation is profoundly influenced. There can be adverse effects on the neurological outcome due to the procedure. The two methods are considered equal, but have never been subjected to comparison. The surgery and circulatory changes can have a negative influence on the cerebral outcome .

METHODS: Twenty patients between 18 and 80 yrs randomized either to crash cooling or gradient cooling, ten patients in each group.. Patients with severe comorbidities or known coagulopathy are excluded. Anesthesia and operation as performed routinely in the department. The primary endpoint is duration of cooling, secondary endpoints include coagulation parameters (thromboelastography, clot stability), stress response parameters (adhesion molecule expression on endothelial cells, oxidative stress analysis, inflammatory markers), neuropsychological tests, MRI of the cerebrum, markers of cerebral ischemia, and ultrasound imaging of the great vessels for detection of air bubbles. Baseline values are obtained for all parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery on the ascending aorta
* Need for deep hypothermic circulatory arrest during the procedure

Exclusion Criteria:

* Known coagulopathy
* Ejection fraction less than 30 %
* Severe psychiatric or neurological disease
* Severe liver disease
* Severely reduced lung function
* Glomerular filtration rate less than 15 ml/min/1.73 m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic. Patients eligible for planned ascending aorta aneurism repair under deep hypothermic circulatory arrest.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Duration of cooling | intraoperatively

SECONDARY OUTCOMES:
MRI of cerebrum | Baseline prior to surgery and 4 to 5 days postoperatively
  Standard perfusion-weighed Magnetic Resonance imaging of the cerebrum. The same investigator describes all images. No use of contrast agents.
Markers of neurological injury | baseline, postoperative
  s-100b, Neuron specific enolase
neurological exam | baseline, postoperative, after 4 months
cognitive test | baseline, postoperative, after 4 months
markers of elevated inflammatory response | perioperatively
Markers of oxidative stress | perioperatively
Coagulation parameters | perioperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anesthesia and intensive care, Aarhus University Hospital, Skejby, Aarhus, Aarhus N, Denmark